CLINICAL TRIAL: NCT02565550
Title: Is Microbiota Community Associated With Clinical Response to a Low FODMAP Diet in Patients With Irritable Bowel Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of Qilu Hospital, Shandong University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015SDU-QILU-G10
Record Dates: First submitted 2015-09-30; First posted 2015-10-01 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Irritable Bowel Syndrome
Keywords: Microbiota Community; FODMAPs; IBS
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — FODMAP Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IBS patients (Experimental): eat the low FODMAPs diet for one week
  Interventions: Dietary Supplement: low FODMAPs
- healthy controls (Active Comparator): eat the low FODMAPs diet for one week
  Interventions: Dietary Supplement: low FODMAPs

INTERVENTIONS:
Dietary Supplement: low FODMAPs — low FODMAPs means excluding food which contains oligosaccharides.disaccharides,monosaccharides, and polyols

SUMMARY:
To determine the efficacy of a low FODMAP diet in IBS patients and whether gut microbiota community is associated with its efficacy.

DETAILED DESCRIPTION:
We seek to determine whether a low FODMAPs diet decreases symptoms in irritable bowel syndrome (IBS)patients and to identify potential microbial factors related to diet efficacy. Pain symptoms, stooling characteristics, breath hydrogen, stool microbiome will be collected and/or documented in IBS patients at baseline and during one week of an low FODMAPs intervention.

ELIGIBILITY:
Inclusion Criteria:

* the presence of Rome III criteria for IBS ;
* Patients scheduled for colonoscopy examination or having negative screening examinations
* Aged between 18 and 65 years old

Exclusion Criteria:

* Antibiotic, probiotic or laxative usage within 4 weeks.
* organic gastrointestinal diseases
* Severe systematic disease: diabetes mellitus, hepatic, renal or cardiac dysfunction, thyroid disease or tumor etc.
* pregnancy or lactation.
* previous major or complicated abdominal surgery.
* severe endometriosis and dementia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-07; Primary Completion 2015-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
changes of symptom scores | 5 months

SECONDARY OUTCOMES:
proportion of responders | 3 months
quality of life in IBS patients | 5 months
microbial composition in different response to low FODMAPs | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, MD.PhD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China